CLINICAL TRIAL: NCT02874326
Title: An Uncontrolled, Pilot-study Assessing the Efficacy of Octreotide Long-acting Release to Decrease Transfusion Requirements and Endoscopy Frequency in Patients With Rendu-Osler-Weber and Gastrointestinal Bleeding
Brief Title: Octreotide in Patients With GI Bleeding Due to Rendu-Osler-Weber
Acronym: ROW
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: St. Antonius Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLROW.1012.15
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Hereditary Hemorrhagic Telangiectasia; Gastrointestinal Hemorrhage; Anemia
Keywords: Sandostatin LAR; Somatostatin; Octreotide
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Gastrointestinal Hemorrhage; Anemia | interventions — Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active comparator: Octreotide LAR (Experimental): Sandostatin LAR Sandostatin LAR 20 mg will be administered once every 4 weeks as a intramuscular injection
  Interventions: Drug: Octreotide LAR

INTERVENTIONS:
Drug: Octreotide LAR
  Other Names: Sandostatin; Dutch registration number (RVG) 18236; Anatomical Therapeutic Chemical (ATC) H01CB02

SUMMARY:
The purpose of this study is to determine whether long-acting octreotide is safe and effective in the treatment of patients with Rendu-Osler-Weber (e.g. HHT).

The study hypothesis is that octreotide is safe and will reduce transfusion requirements and endoscopy frequency in ROW patients with refractory anaemia due to bleeding gastrointestinal telangiectasias.

DETAILED DESCRIPTION:
Rationale: Rendu-Osler-Weber (ROW) is an autosomal dominant hereditary disease which affects 1 / 5-8000 individuals. It is characterized by arteriovenous malformations (AVMs) and telangiectasias in multiple organs, including the gastrointestinal tract. Patients can be transfusion dependent due to severe gastrointestinal bleeding from those telangiectasias. Endoscopy is not as effective due to the recurrent character of the telangiectasias. Based on literature in patients with non-ROW AVMs and telangiectasias, octreotide might be beneficial for these patients to decrease their transfusion needs.

Objective: To assess the efficacy of octreotide in decreasing the need for transfusions and endoscopic intervention in patients ROW with refractory anaemia due to gastrointestinal bleeding telangiectasias.

Study design: Multicenter, open-label uncontrolled pilot study.

Study population: Patients with ROW and symptomatic gastrointestinal bleeding telangiectasias, who are transfusion and/or endoscopy dependent:

1. Transfusion dependent: at least 2 blood and/or iron infusions in the 6 months before inclusion.
2. Endoscopy dependent: at least one endoscopic intervention with argon plasma coagulation (APC) after the initial/first endoscopic treatment after diagnosis in the half year before inclusion or unsuitable for endoscopy.

Intervention: The intervention is 20 mg Sandostatin long-acting release (LAR) once every four weeks for 26 weeks on top of standard of care.

Main study parameters/endpoints: Primary outcome is response to treatment defined as:

* complete: no endoscopic intervention or transfusion requirements
* partial: a reduction in endoscopic intervention or transfusion requirements
* non-response: an equal or increase in endoscopy frequency or transfusions Important secondary outcomes are the percent change in the number of rebleeds from baseline to endpoint and the number of epistaxis episodes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Rendu-Osler-Weber
* Symptomatic gastrointestinal bleeds out of telangiectasias
* Transfusion and / or endoscopy dependent:

Transfusion: at least 2 blood and/or iron infusions in the 6 months before inclusion.

Endoscopy: at least one endoscopy with APC after the initial endoscopic treatment after diagnosis in the half year before inclusion or unsuitable for endoscopic therapy.

Exclusion Criteria:

* liver cirrhosis Child-Pugh C or acute liver failure
* previous unsuccessful treatment with somatostatin analogues (SST) for the same indication (refractory anaemia due to telangiectasias) or current effective treatment with a somatostatin analogue
* severe diseases with life expectancy < 1 year
* patients with left ventricular assist devices (LVAD's)
* Symptomatic cholecystolithiasis (without cholecystectomy)
* pregnancy or nursing women or women who have a pregnancy wish in the study period or who use anticonception inadequate
* current chemotherapy
* patients with a known hypersensitivity to SST analogues or any component of the octreotide LAR formulations
* no understanding of Dutch or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients who are full responder, partial responder and non-responder at the end of the treatment period | Comparing the 6 months before inclusion and the study period (26 weeks)
  Full responder: no endoscopy and no blood/iron transfusions during treatment period.
  * Partial responder: a decrease in number of blood/iron transfusions and/or endoscopy during the treatment period compared with the 6 months prior to inclusion.
  * Non-responder: no decrease in number of blood/iron transfusions and endoscopy during the treatment period compared with the 6 months prior to inclusion.

SECONDARY OUTCOMES:
The percentual decrease in blood and iron requirements | Comparing the 6 months prior to inclusion and the treatment period of 6 months.
The percentual decrease in the number of endoscopic interventions | Comparing the 6 months prior to inclusion and the treatment period of 6 months.
The mean/median decrease on the epistaxis severity score (ESS) | Comparing the 6 months prior to inclusion and the treatment period of 6 months.
  Comparing baseline and the end of treatment visit (week 26)
Change in quality of life using the Short Form (SF)-36 questionnaire | Comparing baseline and end of treatment visit
The number, type and severity of adverse events | Study period

CONTACTS AND LOCATIONS:
Overall Officials: Joost Drenth, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Radboudumc, Nijmegen, Gelderland
  - St Antonius Hospital, Nieuwegein, Utrecht

IPD SHARING:
Plan to Share IPD: No